CLINICAL TRIAL: NCT01216163
Title: Evaluation Of The Efficacy Of A Novel Ibuprofen Formulation In The Treatment Of Post-Surgical Dental Pain
Brief Title: Study Evaluating A Novel Ibuprofen Formulation In The Treatment Of Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-09-14; B3411002
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Pain
Keywords: Pain following third molar extraction (wisdom tooth)
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Novel Ibuprofen
- Treatment B (Active Comparator)
  Interventions: Drug: Acetaminophen
- Treatment C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Novel Ibuprofen — Single-dose of novel ibuprofen (equal to 400 mg ibuprofen)
  Arms: Treatment A
Drug: Acetaminophen — Single-dose of acetaminophen (1000mg)
  Arms: Treatment B
Drug: Placebo — Single-dose of placebo
  Arms: Treatment C

SUMMARY:
This study will compare the analgesic efficacy of a single-dose of a novel ibuprofen formulation to placebo and acetaminophen in the treatment of post-surgical dental pain following "wisdom" tooth (third molar) removal.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy males and females 16 to 40 years of age
* Outpatients who have moderate to severe post-operative pain (confirmed by a Visual Analog Scale-Pain Severity Rating [VAS-PSR] score of at least 50 mm on a 100 mm VAS PSR) following surgical extraction of two or more third molars, at least one of which must be a partial or complete bony mandibular impaction
* Use of only the following pre-operative medication(s)/anesthetic(s): topical benzocaine, a short acting parenteral (local) anesthetic (mepivacaine or lidocaine) with or without vasoconstrictor and/or nitrous oxide

Exclusion Criteria:

* Pregnancy or breast-feeding
* Alcohol or substance abuse
* Any serious medical or psychiatric disorder
* History of stomach ulcers, stomach bleed, or other bleeding disorders
* Use of a prescription or over-the-counter (OTC) drug with which administration of ibuprofen or any other non-steroidal anti-inflammatory drug (NSAID); acetaminophen (APAP); or codeine or any other opioid is contraindicated (including: opioids, antipsychotics, antianxiety agents, or other central nervous system depressants [including alcohol])

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 218 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Jayawardena S, Leyva R, Kellstein D. Safety of a novel formulation of ibuprofen sodium compared with standard ibuprofen and placebo. Postgrad Med. 2015 Jan;127(1):33-7. doi: 10.1080/00325481.2015.993268. Epub 2014 Dec 15. PMID 25526232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3411002&StudyName=Study%20Evaluating%20A%20Novel%20Ibuprofen%20Formulation%20In%20The%20Treatment%20Of%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 milligram (mg) tablet.
- Ibuprofen Sodium: Single oral dose of 2 ibuprofen sodium 256 mg tablets, equivalent to 400 mg ibuprofen.
- Acetaminophen: Single oral dose of 2 acetaminophen (Extra Strength Tylenol) 500 mg tablets, equivalent to 1000 mg acetaminophen.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Started | 45 | 88 | 85
Completed | 44 | 87 | 85
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen | Total
Number analyzed (Participants) | 45 | 88 | 85 | 218
Age Continuous [Mean (Standard Deviation); unit: years] | 19.2 (2.1) | 19.2 (2.8) | 19.1 (2.5) | 19.2 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 45 | 42 | 110
  Male | 22 | 43 | 43 | 108
Number of Participants with Pain Severity Score [Number; unit: participants] — Pain severity score was assessed on a 4-point categorical scale. Total possible pain severity score range was 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
  participants
    Moderate | 33 | 64 | 60 | 157
    Severe | 12 | 24 | 25 | 61

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief Rating With Pain Intensity Difference From 0 to 6 Hours (SPRID 0-6)
Description: SPRID: time-weighted sum of pain relief rating combined with pain intensity difference (PRID) over 6 hours. Score range: -6(worst) to 42(best) for SPRID 0-6. PRID: sum of pain intensity difference (PID) and pain relief rating (PRR) at each time point. Score range for PRID: -1(worst) to 7(best). PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). Total score range for PID: -1 (worst) to 3 (best). PRR: assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 6 hours
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale | 2.8 (9.9) | 20.0 (11.6) | 17.1 (11.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference(Ibuprofen sodium - placebo) and 95 percent(%) confidence interval(CI):based on LS means from Analysis of Variance(ANOVA).Type I error controlled at 5% significance level(2-sided) by testing co-primary endpoints sequentially:Ibuprofen sodium(IBU Na) versus(vs) Placebo(PBO), IBU Na vs Acetaminophen(APAP), APAP vs PBO for SPRID 0-6 then time to meaningful relief at each comparison.If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline Pain Severity Rating (PSR), gender and treatment-by-baseline PSR terms; Least-squares (LS) mean difference = 17.68, 95% CI 2-sided [13.08 to 22.27]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; Treatment difference (Ibuprofen sodium - Acetaminophen) and 95% CI: based on LS means from ANOVA. Type I error controlled at 5% significance level(2-sided) by testing co-primary endpoints sequentially:IBU Na vs PBO, IBU Na vs APAP, APAP vs PBO for SPRID 0-6 then time to meaningful relief at each comparison.If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p = 0.010, ANOVA — p-value was calculated using ANOVA model with treatment, baseline PSR, gender and treatment-by-baseline PSR terms; LS mean difference = 4.96, 95% CI 2-sided [1.21 to 8.72]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; Treatment difference (Acetaminophen - Placebo) and 95% CI: based on LS means from ANOVA. Type I error controlled at 5% significance level(2-sided) by testing co-primary endpoints sequentially:IBU Na vs PBO, IBU Na vs APAP, APAP vs PBO for SPRID 0-6 then time to meaningful relief at each comparison.If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline PSR, gender and treatment-by-baseline PSR terms; LS mean difference = 12.71, 95% CI 2-sided [8.12 to 17.30]

2. Primary Outcome: Time to Onset of Meaningful Relief
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment they first began to experience meaningful relief. Stopwatch was active up to 6 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
minutes | NA [NA to NA] — Data was not summarized as median time to meaningful effect was greater than (>) 360 minutes for Placebo group and therefore 95% CI was not estimable. | 58.0 [41.4 to 74.8] | 53.4 [48.6 to 69.1]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Hazard Ratio (HR) and corresponding 95% CI were calculated based on the Wald statistic from the proportional hazards (PH) model. Type I error controlled at 5% significance level(2-sided) by testing co-primary endpoints sequentially:IBU Na vs PBO, IBU Na vs APAP, APAP vs PBO for SPRID 0-6 then time to meaningful relief at each comparison.If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms; Hazard Ratio (HR) = 11.84, 95% CI 2-sided [5.13 to 27.36]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model. Type I error controlled at 5% significance level(2-sided) by testing co-primary endpoints sequentially:IBU Na vs PBO, IBU Na vs APAP, APAP vs PBO for SPRID 0-6 then time to meaningful relief at each comparison.If comparison at preceding step was significant only then subsequent comparisons were significant; Test type: Superiority or Other; p = 0.468, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.81 to 1.60]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms; Hazard Ratio (HR) = 10.43, 95% CI 2-sided [4.50 to 24.17]

3. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment they first began to experience any relief. Stopwatch was active up to 6 hours after dosing or until stopped by the participant, or rescue medication was administered. The first perceptible relief was considered confirmed if the participant also stopped the second stopwatch indicating meaningful relief.
Time Frame: 0 to 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
minutes | NA [NA to NA] — Data was not summarized as median time to first confirmed perceptible relief was >360 minutes for Placebo group and therefore 95% CI was not estimable. | 16.0 [15.7 to 26.8] | 23.7 [19.0 to 29.3]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 14.06, 95% CI 2-sided [6.02 to 32.80]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.323, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.84 to 1.68]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 11.81, 95% CI 2-sided [5.06 to 27.59]

4. Secondary Outcome: Pain Relief Rating (PRR)
Description: PRR was evaluated at different time points during the study up to 6 hours after taking the study medication, and immediately before rescue medication was taken (if necessary). PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  0.25 hours | 0.1 (0.4) | 0.7 (0.8) | 0.4 (0.7)
  0.5 hours | 0.3 (0.6) | 1.8 (1.2) | 1.5 (1.1)
  1 hour | 0.6 (0.8) | 2.6 (1.1) | 2.4 (1.2)
  1.5 hours | 0.5 (0.9) | 2.8 (1.1) | 2.5 (1.2)
  2 hours | 0.5 (1.1) | 2.8 (1.2) | 2.5 (1.4)
  3 hours | 0.5 (1.1) | 2.5 (1.4) | 2.2 (1.5)
  4 hours | 0.5 (1.2) | 2.4 (1.5) | 2.1 (1.6)
  5 hours | 0.5 (1.2) | 2.0 (1.5) | 1.9 (1.6)
  6 hours | 0.5 (1.2) | 2.0 (1.6) | 1.7 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline PSR, gender and treatment-by-baseline PSR terms. Statistical testing was done at 5% significance level (2-sided); LS mean difference = 0.53, 95% CI 2-sided [0.24 to 0.83]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; 0.25 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.101, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.20, 95% CI 2-sided [-0.04 to 0.44]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; 0.25 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.029, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.33, 95% CI 2-sided [0.03 to 0.62]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.44, 95% CI 2-sided [1.01 to 1.87]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; 0.5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.178, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.24, 95% CI 2-sided [-0.11 to 0.59]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; 0.5 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.20, 95% CI 2-sided [0.77 to 1.63]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.07, 95% CI 2-sided [1.64 to 2.49]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; 1 hour: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.014, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.44, 95% CI 2-sided [0.09 to 0.78]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; 1 hour: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.63, 95% CI 2-sided [1.21 to 2.06]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; 1.5 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.25, 95% CI 2-sided [1.79 to 2.70]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; 1.5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.055, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.37, 95% CI 2-sided [-0.01 to 0.74]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; 1.5 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.88, 95% CI 2-sided [1.43 to 2.34]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.31, 95% CI 2-sided [1.80 to 2.83]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; 2 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.019, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.51, 95% CI 2-sided [0.08 to 0.93]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; 2 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.81, 95% CI 2-sided [1.29 to 2.32]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.10, 95% CI 2-sided [1.53 to 2.66]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; 3 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.013, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.59, 95% CI 2-sided [0.13 to 1.05]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; 3 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.51, 95% CI 2-sided [0.95 to 2.07]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.97, 95% CI 2-sided [1.39 to 2.56]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Acetaminophen; 4 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.63, 95% CI 2-sided [0.15 to 1.10]
Statistical Analysis 21: Comparison: Placebo vs Acetaminophen; 4 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.35, 95% CI 2-sided [0.77 to 1.93]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen Sodium; 5 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.54, 95% CI 2-sided [0.95 to 2.14]
Statistical Analysis 23: Comparison: Ibuprofen Sodium vs Acetaminophen; 5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.088, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.42, 95% CI 2-sided [-0.06 to 0.91]
Statistical Analysis 24: Comparison: Placebo vs Acetaminophen; 5 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.12, 95% CI 2-sided [0.52 to 1.71]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.46, 95% CI 2-sided [0.85 to 2.07]
Statistical Analysis 26: Comparison: Ibuprofen Sodium vs Acetaminophen; 6 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.061, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.47, 95% CI 2-sided [-0.02 to 0.97]
Statistical Analysis 27: Comparison: Placebo vs Acetaminophen; 6 hours: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.98, 95% CI 2-sided [0.38 to 1.59]

5. Secondary Outcome: Pain Intensity Difference (PID)
Description: PID was derived by subtracting the pain severity score at a given post-dosing time point (pain severity score range 0 [none] to 3 [severe]) from the baseline score (Baseline pain severity score range 2 [moderate] to 3 [severe]). Total possible score range for PID: -1 (worst) to 3 (best).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  0.25 hours | -0.1 (0.3) | 0.3 (0.5) | 0.2 (0.5)
  0.5 hours | -0.1 (0.4) | 0.8 (0.7) | 0.5 (0.7)
  1 hour | 0.0 (0.6) | 1.3 (0.8) | 1.0 (0.8)
  1.5 hours | -0.0 (0.7) | 1.3 (0.8) | 1.1 (0.9)
  2 hours | -0.0 (0.8) | 1.3 (0.9) | 1.1 (1.0)
  3 hours | -0.0 (0.9) | 1.2 (1.0) | 0.9 (0.9)
  4 hours | -0.0 (0.8) | 1.1 (1.0) | 0.9 (0.9)
  5 hours | 0.0 (0.9) | 0.9 (1.0) | 0.8 (0.9)
  6 hours | -0.0 (0.9) | 0.9 (1.1) | 0.6 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.31, 95% CI 2-sided [0.13 to 0.49]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.387, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.06, 95% CI 2-sided [-0.08 to 0.21]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [0.07 to 0.42]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.89, 95% CI 2-sided [0.64 to 1.15]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.019, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [0.04 to 0.46]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.64, 95% CI 2-sided [0.38 to 0.90]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.30, 95% CI 2-sided [1.01 to 1.59]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.33, 95% CI 2-sided [0.09 to 0.57]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.97, 95% CI 2-sided [0.68 to 1.26]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.43, 95% CI 2-sided [1.12 to 1.74]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.014, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.32, 95% CI 2-sided [0.07 to 0.58]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.11, 95% CI 2-sided [0.80 to 1.42]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.43, 95% CI 2-sided [1.09 to 1.78]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 14]; Test type: Superiority or Other; p = 0.030, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.31, 95% CI 2-sided [0.03 to 0.59]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.12, 95% CI 2-sided [0.78 to 1.46]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.29, 95% CI 2-sided [0.91 to 1.66]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.42, 95% CI 2-sided [0.12 to 0.73]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 18]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.87, 95% CI 2-sided [0.49 to 1.24]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.27, 95% CI 2-sided [0.89 to 1.65]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 20]; Test type: Superiority or Other; p = 0.004, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.45, 95% CI 2-sided [0.15 to 0.76]
Statistical Analysis 21: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.82, 95% CI 2-sided [0.44 to 1.19]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.92, 95% CI 2-sided [0.54 to 1.31]
Statistical Analysis 23: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 23]; Test type: Superiority or Other; p = 0.084, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.28, 95% CI 2-sided [-0.04 to 0.59]
Statistical Analysis 24: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 24]; Test type: Superiority or Other; p = 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.65, 95% CI 2-sided [0.27 to 1.03]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.93, 95% CI 2-sided [0.54 to 1.32]
Statistical Analysis 26: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.020, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.38, 95% CI 2-sided [0.06 to 0.69]
Statistical Analysis 27: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 27]; Test type: Superiority or Other; p = 0.005, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.56, 95% CI 2-sided [0.17 to 0.94]

6. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference (PRID)
Description: PRID was sum of PID and PRR at each post-dosing time point. The overall possible score range, for PRID was -1 (worst) to 7 (best). PID was derived by subtracting the pain severity score at a given post-dosing time point (pain severity score range 0 [none] to 3 [severe]) from the baseline score (Baseline pain severity score range 2 [moderate] to 3 [severe]). Total possible score range for PID: -1 (worst) to 3 (best). PRR was assessed on 5-point categorical pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  0.25 hours | 0.1 (0.5) | 0.9 (1.3) | 0.6 (1.1)
  0.5 hours | 0.2 (0.8) | 2.5 (1.8) | 2.0 (1.7)
  1 hour | 0.6 (1.3) | 3.9 (1.8) | 3.4 (1.9)
  1.5 hours | 0.5 (1.5) | 4.1 (1.9) | 3.7 (2.0)
  2 hours | 0.5 (1.8) | 4.1 (2.0) | 3.6 (2.3)
  3 hours | 0.4 (1.9) | 3.7 (2.3) | 3.1 (2.4)
  4 hours | 0.5 (1.9) | 3.6 (2.4) | 3.0 (2.4)
  5 hours | 0.5 (2.1) | 2.9 (2.5) | 2.7 (2.5)
  6 hours | 0.5 (1.9) | 2.8 (2.6) | 2.3 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.84, 95% CI 2-sided [0.40 to 1.28]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.148, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.27, 95% CI 2-sided [-0.10 to 0.63]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.011, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.57, 95% CI 2-sided [0.13 to 1.02]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.34, 95% CI 2-sided [1.68 to 2.99]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.071, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.49, 95% CI 2-sided [-0.04 to 1.03]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.84, 95% CI 2-sided [1.19 to 2.50]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.37, 95% CI 2-sided [2.67 to 4.06]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.008, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.77, 95% CI 2-sided [0.20 to 1.33]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.60, 95% CI 2-sided [1.91 to 3.30]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.68, 95% CI 2-sided [2.92 to 4.43]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.028, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.69, 95% CI 2-sided [0.07 to 1.30]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.99, 95% CI 2-sided [2.24 to 3.74]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.75, 95% CI 2-sided [2.90 to 4.59]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 14]; Test type: Superiority or Other; p = 0.020, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.82, 95% CI 2-sided [0.13 to 1.51]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.93, 95% CI 2-sided [2.09 to 3.77]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.38, 95% CI 2-sided [2.46 to 4.30]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.009, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.01, 95% CI 2-sided [0.26 to 1.76]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 18]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.38, 95% CI 2-sided [1.46 to 3.30]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.24, 95% CI 2-sided [2.30 to 4.19]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 20]; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.08, 95% CI 2-sided [0.31 to 1.85]
Statistical Analysis 21: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.16, 95% CI 2-sided [1.22 to 3.10]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.47, 95% CI 2-sided [1.51 to 3.43]
Statistical Analysis 23: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 23]; Test type: Superiority or Other; p = 0.080, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.70, 95% CI 2-sided [-0.09 to 1.49]
Statistical Analysis 24: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 24]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.77, 95% CI 2-sided [0.81 to 2.73]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.39, 95% CI 2-sided [1.41 to 3.37]
Statistical Analysis 26: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.037, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.85, 95% CI 2-sided [0.05 to 1.65]
Statistical Analysis 27: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 4, analysis 27]; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.54, 95% CI 2-sided [0.57 to 2.52]

7. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID)
Description: SPID: time-weighted sum of PID over 2, 3 and 6 hours. Total score range: -2 (worst) to 6 (best) for SPID 0-2, -3 (worst) to 9 (best) for SPID 0-3, and -6 (worst) to 18 (best) for SPID 0-6. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). Total score range for PID: -1 (worst) to 3 (best).
Time Frame: 0 to 2, 0 to 3, 0 to 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  SPID 0-2 | -0.1 (1.1) | 2.2 (1.4) | 1.8 (1.4)
  SPID 0-3 | -0.1 (1.9) | 3.4 (2.3) | 2.8 (2.1)
  SPID 0-6 | -0.1 (4.4) | 6.3 (5.0) | 5.1 (4.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-2: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.38, 95% CI 2-sided [1.88 to 2.88]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; SPID 0-2: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.56, 95% CI 2-sided [0.15 to 0.97]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; SPID 0-2: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.82, 95% CI 2-sided [1.32 to 2.32]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-3: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.67, 95% CI 2-sided [2.85 to 4.49]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; SPID 0-3: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.004, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.98, 95% CI 2-sided [0.31 to 1.66]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; SPID 0-3: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.69, 95% CI 2-sided [1.87 to 3.51]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-6: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 6.80, 95% CI 2-sided [4.96 to 8.64]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; SPID 0-6: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.09, 95% CI 2-sided [0.59 to 3.59]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; SPID 0-6: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.71, 95% CI 2-sided [2.87 to 6.54]

8. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR)
Description: TOTPAR: time-weighted sum of PRR over 2, 3, and 6 hours. Total score range: 0 (worst) to 8 (best) for TOTPAR 0-2, 0 (worst) to 12 (best) for TOTPAR 0-3, and 0 (worst) to 24 (best) for TOTPAR 0-6. PRR was evaluated at different time points during the study up to 6 hours, and immediately after taking rescue medication (if necessary). PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 0 to 2, 0 to 3, 0 to 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  TOTPAR 0-2 | 0.9 (1.4) | 4.7 (1.9) | 4.2 (2.0)
  TOTPAR 0-3 | 1.4 (2.5) | 7.2 (3.1) | 6.4 (3.4)
  TOTPAR 0-6 | 2.9 (5.9) | 13.6 (7.0) | 12.0 (7.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-2: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.81, 95% CI 2-sided [3.05 to 4.57]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; TOTPAR 0-2: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.016, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 0.76, 95% CI 2-sided [0.14 to 1.38]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; TOTPAR 0-2: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 3.04, 95% CI 2-sided [2.29 to 3.80]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-3: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 5.90, 95% CI 2-sided [4.66 to 7.15]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; TOTPAR 0-3: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.35, 95% CI 2-sided [0.33 to 2.37]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; TOTPAR 0-3: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.56, 95% CI 2-sided [3.31 to 5.80]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-6: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 10.88, 95% CI 2-sided [8.05 to 13.70]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; TOTPAR 0-6: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.015, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.87, 95% CI 2-sided [0.57 to 5.18]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; TOTPAR 0-6: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 8.00, 95% CI 2-sided [5.18 to 10.83]

9. Secondary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference (SPRID)
Description: SPRID: time-weighted sum of PRID over 2 and 3 hours. Total score range: -2 (worst) to 14 (best) for SPRID 0-2, and -3 (worst) to 21 (best) for SPRID 0-3. PRID: sum of PID and PRR at each time point. Total score range for PRID: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderate to 3=severe). Total score range for PID: -1 (worst) to 3 (best). PRR: assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale
  SPRID 0-2 | 0.9 (2.4) | 6.9 (3.1) | 6.0 (3.3)
  SPRID 0-3 | 1.3 (4.2) | 10.6 (5.2) | 9.1 (5.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-2: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 6.19, 95% CI 2-sided [4.96 to 7.43]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; SPRID 0-2: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 1.33, 95% CI 2-sided [0.32 to 2.33]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; SPRID 0-2: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 4.87, 95% CI 2-sided [3.63 to 6.10]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-3: Treatment difference (Ibuprofen sodium - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 9.58, 95% CI 2-sided [7.54 to 11.61]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; SPRID 0-3: Treatment difference (Ibuprofen sodium - Acetaminophen) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.33, 95% CI 2-sided [0.67 to 4.00]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; SPRID 0-3: Treatment difference (Acetaminophen - Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 7.24, 95% CI 2-sided [5.21 to 9.28]

10. Secondary Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief evaluated by stopping the stopwatch labeled 'meaningful relief' at the moment participant first began to experience meaningful relief. Stopwatch was active up to 6 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
percentage of participants
  0.25 hours | 0.0 | 0.0 | 0.0
  0.5 hours | 0.0 | 21.6 | 20.0
  1 hour | 0.0 | 53.4 | 56.5
  1.5 hours | 2.2 | 72.7 | 64.7
  2 hours | 8.9 | 75.0 | 70.6
  3 hours | 11.1 | 77.3 | 71.8
  4 hours | 13.3 | 78.4 | 74.1
  5 hours | 13.3 | 79.5 | 74.1
  6 hours | 13.3 | 79.5 | 74.1
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value was calculated using CMH test, controlling for baseline PSR and gender. Statistical testing was done at 5% significance level (2-sided); Difference in proportion = 21.42, 95% CI 2-sided [12.99 to 29.84]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; 0.5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.799, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.58, 95% CI 2-sided [-10.54 to 13.70]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; 0.5 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 20.09, 95% CI 2-sided [11.45 to 28.72]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 53.22, 95% CI 2-sided [42.92 to 63.53]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; 1 hour: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.695, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -2.98, 95% CI 2-sided [-17.67 to 11.70]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; 1 hour: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 57.06, 95% CI 2-sided [46.53 to 67.60]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 1.5 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 70.58, 95% CI 2-sided [60.28 to 80.88]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; 1.5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.261, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 7.99, 95% CI 2-sided [-5.85 to 21.84]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; 1.5 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 62.88, 95% CI 2-sided [51.78 to 73.99]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.24, 95% CI 2-sided [53.77 to 78.71]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; 2 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.522, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 4.38, 95% CI 2-sided [-8.89 to 17.64]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; 2 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.93, 95% CI 2-sided [49.06 to 74.80]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.35, 95% CI 2-sided [53.61 to 79.09]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; 3 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.415, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.46, 95% CI 2-sided [-7.53 to 18.44]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; 3 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 60.92, 95% CI 2-sided [47.65 to 74.19]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 65.32, 95% CI 2-sided [52.18 to 78.46]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; 4 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.519, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 4.21, 95% CI 2-sided [-8.39 to 16.81]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; 4 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; 5 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Acetaminophen; 5 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 21: Comparison: Placebo vs Acetaminophen; 5 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 23: Comparison: Ibuprofen Sodium vs Acetaminophen; 6 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 24: Comparison: Placebo vs Acetaminophen; 6 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]

11. Secondary Outcome: Cumulative Percentage of Participants With Confirmed First Perceptible Relief
Description: Percentage of participants with first perceptible relief evaluated by stopping the stopwatch labeled 'first perceptible relief' at the moment participant first began to experience any relief. First perceptible relief was considered confirmed if the participant also stopped the second stopwatch indicating meaningful relief. Stopwatch was active up to 6 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
percentage of participants
  0.25 hours | 2.2 | 28.4 | 24.7
  0.5 hours | 4.4 | 64.8 | 62.4
  1 hour | 11.1 | 78.4 | 72.9
  1.5 hours | 11.1 | 79.5 | 74.1
  2 hours | 13.3 | 79.5 | 74.1
  3 hours | 13.3 | 79.5 | 74.1
  4 hours | 13.3 | 79.5 | 74.1
  5 hours | 13.3 | 79.5 | 74.1
  6 hours | 13.3 | 79.5 | 74.1
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 26.40, 95% CI 2-sided [15.87 to 36.93]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; 0.25 hours: Treatment difference (Ibuprofen sodium - Acetaminophen) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.602, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 3.53, 95% CI 2-sided [-9.85 to 16.91]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; 0.25 hours: Treatment difference (Acetaminophen - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 22.72, 95% CI 2-sided [12.39 to 33.05]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - Placebo) and its associated CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 60.37, 95% CI 2-sided [48.61 to 72.12]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.761, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 2.25, 95% CI 2-sided [-12.10 to 16.59]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 58.32, 95% CI 2-sided [46.59 to 70.05]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 67.52, 95% CI 2-sided [54.91 to 80.12]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.410, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.42, 95% CI 2-sided [-7.34 to 18.18]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 62.13, 95% CI 2-sided [48.96 to 75.29]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 68.64, 95% CI 2-sided [56.11 to 81.16]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 63.34, 95% CI 2-sided [50.32 to 76.35]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 20: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 21: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 23: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 24: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 66.44, 95% CI 2-sided [53.38 to 79.51]
Statistical Analysis 26: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 23]; Test type: Superiority or Other; p = 0.412, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 5.31, 95% CI 2-sided [-7.22 to 17.83]
Statistical Analysis 27: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 24]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 61.14, 95% CI 2-sided [47.60 to 74.68]

12. Secondary Outcome: Time to Treatment Failure
Description: Median time of dropping out of the participants from the study due to lack of efficacy or use of rescue medication, whichever comes first.
Time Frame: 0 to 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
hours | 1.6 [1.4 to 1.9] | NA [NA to NA] — Data was not summarized as median time to treatment failure was >6 hours for Ibuprofen sodium group and therefore 95% CI was not estimable. | NA [NA to NA] — Data was not summarized as median time to treatment failure was >6 hours for Acetaminophen group and therefore 95% CI was not estimable.
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.08 to 0.22]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.303, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.45 to 1.28]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.10 to 0.28]

13. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Percentage of participants who withdrew from the study due to lack of efficacy or received rescue medication.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
percentage of participants
  0.25 hours | 0.0 | 0.0 | 0.0
  0.5 hours | 0.0 | 0.0 | 0.0
  1 hour | 0.0 | 0.0 | 0.0
  1.5 hours | 42.2 | 2.3 | 2.4
  2 hours | 68.9 | 5.7 | 12.9
  3 hours | 82.2 | 11.4 | 21.2
  4 hours | 82.2 | 15.9 | 27.1
  5 hours | 82.2 | 25.0 | 32.9
  6 hours | 82.2 | 29.5 | 35.3
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -40.10, 95% CI 2-sided [-55.39 to -24.80]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.958, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -0.12, 95% CI 2-sided [-4.52 to 4.28]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -40.19, 95% CI 2-sided [-55.51 to -24.87]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -63.40, 95% CI 2-sided [-77.81 to -48.99]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.108, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -7.17, 95% CI 2-sided [-15.91 to 1.57]
Statistical Analysis 6: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -56.39, 95% CI 2-sided [-71.68 to -41.09]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -71.01, 95% CI 2-sided [-84.09 to -57.93]
Statistical Analysis 8: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.083, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -9.82, 95% CI 2-sided [-20.18 to 1.16]
Statistical Analysis 9: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -61.14, 95% CI 2-sided [-75.40 to -46.87]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -66.37, 95% CI 2-sided [-80.08 to -52.66]
Statistical Analysis 11: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p = 0.079, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -11.03, 95% CI 2-sided [-23.37 to 1.21]
Statistical Analysis 12: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -55.53, 95% CI 2-sided [-70.12 to -40.85]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -57.33, 95% CI 2-sided [-71.90 to -42.77]
Statistical Analysis 14: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.263, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -7.73, 95% CI 2-sided [-21.08 to 5.63]
Statistical Analysis 15: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -49.93, 95% CI 2-sided [-64.74 to -35.12]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -52.75, 95% CI 2-sided [-67.62 to -37.88]
Statistical Analysis 17: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 23]; Test type: Superiority or Other; p = 0.439, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -5.51, 95% CI 2-sided [-19.27 to 8.25]
Statistical Analysis 18: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 24]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -47.72, 95% CI 2-sided [-62.62 to -32.83]

14. Secondary Outcome: Cumulative Percentage of Participants With Complete Relief
Description: Complete relief was defined as a PRR of 4. PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
percentage of participants
  0.25 hours | 0.0 | 0.0 | 1.2
  0.5 hours | 0.0 | 6.8 | 4.7
  1 hours | 0.0 | 23.9 | 15.3
  1.5 hours | 0.0 | 29.5 | 24.7
  2 hours | 4.4 | 36.4 | 29.4
  3 hours | 4.4 | 42.0 | 32.9
  4 hours | 6.7 | 45.5 | 35.3
  5 hours | 8.9 | 45.5 | 35.3
  6 hours | 8.9 | 46.6 | 35.3
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.294, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = -1.21, 95% CI 2-sided [-3.59 to 1.17]
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.458, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.21, 95% CI 2-sided [-1.16 to 3.58]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.81, 95% CI 2-sided [1.57 to 12.06]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.583, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 1.96, 95% CI 2-sided [-4.94 to 8.85]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.137, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 4.81, 95% CI 2-sided [0.14 to 9.49]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 23.86, 95% CI 2-sided [14.81 to 32.91]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.165, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 8.45, 95% CI 2-sided [-3.43 to 20.33]
Statistical Analysis 8: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 15.46, 95% CI 2-sided [7.66 to 23.26]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 29.41, 95% CI 2-sided [19.78 to 39.05]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.497, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 4.61, 95% CI 2-sided [-8.78 to 17.99]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 25.13, 95% CI 2-sided [15.81 to 34.46]
Statistical Analysis 12: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 31.78, 95% CI 2-sided [20.03 to 43.53]
Statistical Analysis 13: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.349, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 6.70, 95% CI 2-sided [-7.38 to 20.79]
Statistical Analysis 14: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 25.34, 95% CI 2-sided [13.73 to 36.94]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 37.64, 95% CI 2-sided [25.47 to 49.81]
Statistical Analysis 16: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.233, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 8.85, 95% CI 2-sided [-5.72 to 23.42]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 28.96, 95% CI 2-sided [17.17 to 40.75]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 38.73, 95% CI 2-sided [25.87 to 51.60]
Statistical Analysis 19: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 17]; Test type: Superiority or Other; p = 0.189, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 9.83, 95% CI 2-sided [-4.80 to 24.45]
Statistical Analysis 20: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 18]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 29.19, 95% CI 2-sided [16.71 to 41.66]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 36.55, 95% CI 2-sided [23.22 to 49.88]
Statistical Analysis 22: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 20]; Test type: Superiority or Other; p = 0.189, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 9.83, 95% CI 2-sided [-4.80 to 24.45]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 21]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 26.97, 95% CI 2-sided [14.00 to 39.94]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 10, analysis 22]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 37.72, 95% CI 2-sided [24.36 to 51.07]
Statistical Analysis 25: Comparison: Ibuprofen Sodium vs Acetaminophen; [analysis description as in outcome 10, analysis 23]; Test type: Superiority or Other; p = 0.144, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 10.97, 95% CI 2-sided [-3.67 to 25.61]
Statistical Analysis 26: Comparison: Placebo vs Acetaminophen; [analysis description as in outcome 10, analysis 24]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Difference in proportion = 26.97, 95% CI 2-sided [14.00 to 39.94]

15. Secondary Outcome: Participant Global Evaluation of Study Medication
Description: Participant global evaluation of study medication was performed at the 6-hour time point or immediately before taking the rescue medication. It was scored on a 6-point categorical scale where 0 = Very poor, 1 = Poor, 2 = Fair, 3 = Good, 4 = Very Good, and 5 = Excellent.
Time Frame: 6 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Number analyzed (Participants) | 45 | 88 | 85
units on a scale | 0.9 (1.3) | 3.5 (1.3) | 3.0 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium - Placebo) and the associated CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test with modified ridit scores, controlling for baseline PSR and gender. Statistical testing was done at 5% significance level (2-sided); Mean Difference (Final Values) = 0.87, 95% CI 2-sided [0.78 to 0.96]
Statistical Analysis 2: Comparison: Ibuprofen Sodium vs Acetaminophen; Treatment difference (Ibuprofen sodium - Acetaminophen) and the associated CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.05 to 0.45]
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen; Treatment difference (Acetaminophen - Placebo) and the associated CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [0.63 to 0.91]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen Sodium | Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/88 | 0/85
Other Adverse Events (participants affected / at risk) | 10/45 | 5/88 | 11/85
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | Ibuprofen Sodium (N=88) | Acetaminophen (N=85)
Dizziness (Nervous system disorders) | 1 | 2 | 5
Headache (Nervous system disorders) | 1 | 1 | 3
Somnolence (Nervous system disorders) | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Hyperhidrosis (General disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.